CLINICAL TRIAL: NCT03098927
Title: Mirror Neuron Network Based Motor Imagery Training Paradigms to Improve Brain Computer Interface (BCI) Performance in Spinal Cord Injury Patients
Brief Title: Mirror Neuron Network Based Motor Imagery Training to Improve Brain Computer Interface Performance in Spinal Cord Injury Patients
Acronym: BCI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Two subjects finally recruited 11/17, but not enough time to complete their studies before the funding terminated on November 30, 2017
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency); MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Hubert Fernandez, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-041
Record Dates: First submitted 2017-03-07; First posted 2017-04-04 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries
Keywords: Motor Imagery; Spinal Cord Injury; Motor Function Improvement
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Eight subjects with spinal cord injury (SCI) will be recruited during the sub-acute phase (3-6 months following injury). Four participants will immediately undergo motor imagery training in an immersive virtual reality environment at NASA. EEG assessments and motor function testing will be performed at intervals during the 3-4 week motor imagery training period to assess improvement in cortical signature generation and motor recovery. The other four participants will undergo the same protocol after a 6 week delay, in order to assess the effect of training timing after injury in both cortical signature generation and motor function recovery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention (Active Comparator): Early intervention patients will undergo 3 weeks of motor imagery training immediately upon enrolling in the study between 3 and 6 months post spinal cord injury.
  Interventions: Behavioral: Motor imagery training
- Late intervention (Active Comparator): Late intervention patients will undergo 3 weeks of motor imagery training after 6 weeks of standard of care physical rehabilitation following enrollment.
  Interventions: Behavioral: Motor imagery training

INTERVENTIONS:
Behavioral: Motor imagery training — Motor imagery training

SUMMARY:
The overall vision of this proposal is to demonstrate that a virtual reality based motor imagery training program will improve brain computer interface (BCI) performance and motor function in quadriplegic subjects. The ultimate goal is to increase the independence of subjects with spinal cord injury by training to safely control BCI assistive devices and to enhance motor recovery.

DETAILED DESCRIPTION:
Intend to train subjects in motor imagery techniques using an advanced virtual reality based platform. Hypothesize that this will enhance the cortical signals necessary for operating a non-invasive EEG-based BCI. Specifically, designed training paradigms will activate "mirror neurons" associated with performance of movement, observation of movement, and motor imagery. Mirror neuron network (MNN) activation induces cortical plasticity, and may therefore enhance cortical signals generated during BCI use. Plan to assess the effect of training paradigm on cortical signals generated during motor imagery, using EEG. Also, investigate neuropsychological factors that play a role in a subject's ability to generate vivid motor imagery.

Eight subjects with spinal cord injury (SCI) will be recruited during the sub-acute phase (3-6 months following injury). Four participants will immediately undergo motor imagery training in an immersive virtual reality environment at NASA. EEG assessments and motor function testing will be performed at intervals during the 3-4 week motor imagery training period to assess improvement in cortical signature generation and motor recovery. The other four participants will undergo the same protocol after a 6 week delay, in order to assess the effect of training timing after injury in both cortical signature generation and motor function recovery.

ELIGIBILITY:
Inclusion Criteria:

* sustained incomplete Spinal Cord Injury (American Spinal Injury Impairment Scale) at a level of C5-7 within three to six months prior to enrollment

Exclusion Criteria:

* unstable or acute medical or psychiatric illness; pregnancy; epilepsy; diabetes; autism spectrum disorder, history of severe traumatic brain injury or stroke, and those taking medications that may interfere with EEG readings, including beta blockers and sedatives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in motor imagery performance | Year 1
  Improvement in scores on Motor Imagery questionnaire
Cortical signal generation (Mirror Neuron Network activation) | Year 2
  EEG collection of cortical activity to quantify changes and discriminate between different types of executed movements during Motor Imagery

CONTACTS AND LOCATIONS:
Overall Officials: Darlene Lobel, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No